CLINICAL TRIAL: NCT00110552
Title: Effects of a Cognitive Enhancer on Memory and Cognitive Performance
Brief Title: Effects of Sage on Memory and Mental Performance in Alzheimer's Disease Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Barry S. Oken, MD, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U19AT002656-03 (NIH); U19AT002656-03 (NIH)
Record Dates: First submitted 2005-05-10; First posted 2005-05-11 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Sage capsules taken by mouth
  Interventions: Drug: Salvia officinalis (sage)
- 2 (No Intervention): No intervention, no-pill as control

INTERVENTIONS:
Drug: Salvia officinalis (sage) — oral dosage
  Other Names: sage
  Arms: 1

SUMMARY:
The purpose of this study is to determine the effectiveness of the herb sage in improving the mental function of individuals with Alzheimer's disease.

Study hypothesis: The administration of sage will improve cognitive function in patients with mild Alzheimer's disease.

DETAILED DESCRIPTION:
The herb sage has been shown to enhance memory and mental function in healthy, young adults. However, studies assessing the herb's effectiveness in older adults with symptoms of Alzheimer's disease are limited. This study will determine the effect of sage extract on the cognitive function of patients with mild Alzheimer's disease.

This study will last 6 weeks and will comprise 4 study visits, approximately 10 days apart. Participants will be randomly assigned to receive either sage pills or no treatment during each 10-day period. The treatment assignments will be switched in 10-day intervals, so that during the course of the study, each participant will undergo two periods of sage treatment and two periods without treatment. At each study visit, participants will undergo cognitive testing, including tests to determine attention, memory, and visual cognition. Participants will also undergo an electroencephalogram (EEG) and an electrocardiogram (ECG) at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild Alzheimer's disease
* Partner, friend, child, spouse, or relative willing to accompany participants to all study visits, provide informed consent, monitor participants' pill-taking, and communicate changes in participants' health during the study

Exclusion Criteria:

* Significant medical illness other than Alzheimer's disease

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2005-07; Primary Completion 2012-12 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Cognitive function | 8 weeks

SECONDARY OUTCOMES:
Stress | 8 weeks
cognitive electrophysiology | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Barry Oken, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Akhondzadeh S, Noroozian M, Mohammadi M, Ohadinia S, Jamshidi AH, Khani M. Salvia officinalis extract in the treatment of patients with mild to moderate Alzheimer's disease: a double blind, randomized and placebo-controlled trial. J Clin Pharm Ther. 2003 Feb;28(1):53-9. doi: 10.1046/j.1365-2710.2003.00463.x. PMID 12605619
- [Background] Perry NS, Bollen C, Perry EK, Ballard C. Salvia for dementia therapy: review of pharmacological activity and pilot tolerability clinical trial. Pharmacol Biochem Behav. 2003 Jun;75(3):651-9. doi: 10.1016/s0091-3057(03)00108-4. PMID 12895683